CLINICAL TRIAL: NCT04388059
Title: Effect of Antrum Size on Glucagon-like Peptide 1 (GLP1) Levels and Glycemic Control After Sleeve Gastrectomy in Morbid Obese Diabetic Adolescents
Brief Title: Antrum Size, Glucagon-like Peptide 1 Levels and Glycemic Control After Sleeve Gastrectomy in Morbid Obese Diabetic Adolescents
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Shehata, Lecturer of pediatric surgery, Tanta University
Other Study IDs: sleeve gastrectomy adolescent
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Adolescent Obesity
Keywords: Laparoscopic sleeve gastrectomy; obesity; adolescent; glucagon-like peptide 1; glycemic control; diabetes
MeSH Terms: conditions — Pediatric Obesity; Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — glucagon-like peptide 1 HbA1c (glycated hemoglobin) body mass index
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transection at 2 cm from the pylorus: the effect of transection at 2 cm from the pylorus during Laparoscopic sleeve gastrectomy on the postoperative weight loss, GLP1 levels and the glycemic control in morbid obese diabetic adolescents.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- Transection at 5 cm from the pylorus: the effect of transection at 5 cm from the pylorus during Laparoscopic sleeve gastrectomy on the postoperative weight loss, GLP1 levels and the glycemic control in morbid obese diabetic adolescents.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Laparoscopic sleeve gastrectomy at 2 and 5 cm from the pylorus on the postoperative weight loss, GLP1 levels and the glycemic control in morbid obese diabetic adolescents.

SUMMARY:
Childhood obesity can adversely affect every organ and often has serious consequences. Compare the effect of transection at 2cm vs at 5cm from the pylorus during laparoscopic sleeve gastrectomy on the postoperative weight loss, glucagon-like peptide 1 levels and the glycemic control in morbid obese diabetic adolescents.

DETAILED DESCRIPTION:
This was a retrospective sub-analysis included 18 type 2 diabetic morbidly obese adolescents of both genders from a larger study (performed on 67 patients between December 2014 and December 2015) conducted at pediatric surgery unit, surgical department, Egypt. They were divided in 2 groups, done by 2 surgeons, group A (8 patients) the first stable line was at 2 cm from the pylorus, and group B (10 patients) at 5 cm from the pylorus.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent, children (more than 12 years or less than 20 years), with BMI of at least 40 kg/m2, or 35 kg/m2 with an associated co-morbidity (e.g. hypertension, diabetes, dyslipidemia, obstructive sleep apnea, left ventricular hypertrophy, nonalcoholic steatohepatitis, orthopedic problems). Those with failure to achieve clinically significant weight loss (10% of baseline body weight) despite strict participation for at least 6 months in a formal weight management program were included in the study.

Exclusion Criteria:

* Adults, children (less than 12 years or more than 20 years) or their family who do not understand risks and benefits of the intervention, adolescents who are not autonomously motivated to consider operation, those have unrealistic expectations for results of the surgical intervention, or their parents, families or patients who cannot strictly comply with the postoperative nutritional recommendations and long-term medical and nutritional monitoring, presence of a medically correctable cause of obesity (relative contraindication), existence of a medical, psychiatric, or cognitive condition as attention deficit hyperkinetic disorders (ADHD) which may impair the ability of patient to assent to surgery or to adhere to postoperative dietary and medication regimen (relative contraindication), illicit substance abuses in preceding year, lactating, pregnant, or plans for pregnancy in upcoming 2 years and patients refuse to participate were excluded.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: morbid obese diabetic adolescents
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
glucagon-like peptide 1 (GLP1) levels in morbid obese diabetic adolescents. | 24 months post-operative
  glucagon-like peptide 1 (GLP1) levels in morbid obese diabetic adolescents after laparoscopic sleeve gastrectomy at 2 and 5 cm from the pylorus
glycemic control in morbid obese diabetic adolescents. | 24 months post-operative
  glycemic control in morbid obese diabetic adolescents after laparoscopic sleeve gastrectomy at 2 and 5 cm from the pylorus

SECONDARY OUTCOMES:
weight loss in morbid obese diabetic adolescents. | 24 months post-operative
  weight loss in morbid obese diabetic adolescents after laparoscopic sleeve gastrectomy at 2 and 5 cm from the pylorus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shehata MA, Elhaddad A, El-Attar AA, Shehata SM. The Effect of Antrum Size on Weight Loss, Glucagon-Like Peptide-1 (GLP-1) Levels, and Glycemic Control Following Laparoscopic Sleeve Gastrectomy in Adolescents with Obesity and Type 2 Diabetes. Obes Surg. 2021 Oct;31(10):4376-4385. doi: 10.1007/s11695-021-05590-9. Epub 2021 Aug 5. PMID 34355337